CLINICAL TRIAL: NCT02438228
Title: Estimation of Cardiac Output by Nine Different Pulse Contour Algorithms Compared With Transpulmonary Thermodilution
Brief Title: Cardiac Output by Nine Different Pulse Contour Algorithms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Ole Broch, MD, MD, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AZ-138
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Cardiac Output
Keywords: cardiac output; transpulmonary thermodilution; pulse contour analysis; G09.330.380.124

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cardiac output measurement (Other)
  Interventions: Other: Cardiac output measurement

INTERVENTIONS:
Other: Cardiac output measurement — Measurement of cardiac output by transpulmonary thermodilution, nine different pulse contour algorithms and esophageal doppler before, during and after a PLR-maneouvre and every 10 minutes before and after cardiopulmonary Bypass.

SUMMARY:
The aim of the present study is to compare accuracy and precision of Cardiac Output (CO) by nine different pulse contour algorithms with transpulmonary thermodilution before and after cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
After induction of anesthesia, a central venous catheter and a transpulmonary thermodilution catheter (Pulsion Medical Systems, Munich, Germany) are introduced in the right internal jugular vein and in the femoral artery, respectively. The thermodilution catheter is connected to a PiCCO2 monitor (Software version 1.3.0.8). Thereafter, placement of an esophageal doppler probe is performed and the probe is connected to a unique Monitoring System (Deltex Medical, Chichester, UK) with nine different pulse contour algorithms. Cardiac Output by esophageal doppler is used to calibrate the nine different pulse contour algorithms.

After induction of anesthesia and establishment of all monitoring devices, a passive leg raising maneouvre (PLR) is performed and hemodynamic variables including CO by transpulmonary thermodilution (COTPTD) and CO by nine different pulse contour algorithms (COX1-9) are recorded before, during and after PLR. Subsequently, measurements of COTPTD and COX1-9 are carried out every 10 minutes until the beginning of CPB. Fifteen minutes after weaning from cardiopulmonary bypass calibration of nine different pulse contour algorithms by esophageal doppler are performed again and measurements of CITPTD and CIPFX are restarted up to the end of the surgical Intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age with a left ventricular ejection fraction ≥ 0.5.
* Patients undergoing coronary artery bypass grafting.

Exclusion Criteria:

* Patients <18 years of age and with a left ventricular ejection fraction ≤0.5 are not considered for the study.
* Emergency procedures and patients with hemodynamic instability requiring continuous pharmacologic support, intracardiac shunts, severe aortic-, tricuspid- or mitral stenosis or insufficiency and mechanical circulatory support were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Accuracy of cardiac output in l/min by nine different pulse contour algorithms compared with transpulmonary thermodilution | After induction of anesthesia until the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Bein, MD, PhD, Principal Investigator — Asklepios Klinik St. Georg
Locations (1):
- Berthold Bein, Hamburg, Hamburg, Germany

REFERENCES:
- [Background] Schloglhofer T, Gilly H, Schima H. Semi-invasive measurement of cardiac output based on pulse contour: a review and analysis. Can J Anaesth. 2014 May;61(5):452-79. doi: 10.1007/s12630-014-0135-8. Epub 2014 Mar 19. PMID 24643474
- [Background] Critchley LA, Lee A, Ho AM. A critical review of the ability of continuous cardiac output monitors to measure trends in cardiac output. Anesth Analg. 2010 Nov;111(5):1180-92. doi: 10.1213/ANE.0b013e3181f08a5b. Epub 2010 Aug 24. PMID 20736431
- [Background] Suehiro K, Tanaka K, Funao T, Matsuura T, Mori T, Nishikawa K. Systemic vascular resistance has an impact on the reliability of the Vigileo-FloTrac system in measuring cardiac output and tracking cardiac output changes. Br J Anaesth. 2013 Aug;111(2):170-7. doi: 10.1093/bja/aet022. Epub 2013 Mar 10. PMID 23479677
- [Background] Smetkin AA, Hussain A, Kuzkov VV, Bjertnaes LJ, Kirov MY. Validation of cardiac output monitoring based on uncalibrated pulse contour analysis vs transpulmonary thermodilution during off-pump coronary artery bypass grafting. Br J Anaesth. 2014 Jun;112(6):1024-31. doi: 10.1093/bja/aet489. Epub 2014 Feb 13. PMID 24531685
- [Background] Huang L, Critchley LA. An assessment of two Doppler-based monitors to track cardiac output changes in anaesthetised patients undergoing major surgery. Anaesth Intensive Care. 2014 Sep;42(5):631-9. doi: 10.1177/0310057X1404200514. PMID 25233178
- [Background] Singer M. Oesophageal Doppler. Curr Opin Crit Care. 2009 Jun;15(3):244-8. doi: 10.1097/MCC.0b013e32832b7083. PMID 19417642
- [Derived] Broch O, Bein B, Gruenewald M, Masing S, Huenges K, Haneya A, Steinfath M, Renner J. Accuracy of Cardiac Output by Nine Different Pulse Contour Algorithms in Cardiac Surgery Patients: A Comparison with Transpulmonary Thermodilution. Biomed Res Int. 2016;2016:3468015. doi: 10.1155/2016/3468015. Epub 2016 Dec 28. PMID 28116294